CLINICAL TRIAL: NCT01570738
Title: Validation of Home Sleep Testing (WP) Compared to an Overnight Sleep Testing in the Sleep Laboratory
Status: Completed | Type: Observational
Sponsor: Itamar-Medical, Israel (Industry)
Responsible Party: Sponsor
Other Study IDs: Carmel-001
Record Dates: First submitted 2012-03-28; First posted 2012-04-04 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-03

CONDITIONS: Sleep Disorders
Keywords: sleep disorders; sleep apnea; ambulatory device; polysomnography; WatchPAT
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Obstructive sleep apnea syndrome (OSAS) is considered to be a major public health problem. The prevalence of OSAS is estimated at 2% and 4% for adult women and men respectively, most of whom are undiagnosed and untreated. The prevalence of snoring in children is high - 5% in the age group of 6 and less and about 1.5% above. The in-lab sleep study using full Polysomnography (PSG) and the manual scoring criteria set by the American Academy of Sleep Medicine was considered the gold standard for OSAS diagnosis. The high cost of in-lab full night PSG, together with long waiting lists for sleep studies, have led to the commonly used procedure of "split-night" for OSAS patients, as well as to the development of a variety of ambulatory sleep study systems. The primary study objective is to compare the efficacy of the WatchPAT (WP), as an ambulatory device for aiding in the diagnosis of sleep disorders for subjects from age 5 to 90, to the manual scoring of the PSG that serves as a "gold standard".

ELIGIBILITY:
Inclusion Criteria:

1. Age between 5-90
2. Subjects that are able to read understand and sign the informed consent form to undergo an overnight sleep study in the clinical sleep laboratory

Exclusion Criteria:

1. Permanent pacemaker.
2. Severe lung disease.
3. Peripheral neuropathy.
4. Finger deformity that precludes adequate sensor appliance.
5. Using one of the following medications: short/Long acting nitrates (less than 3 hours before the sleep study) or alpha-adrenergic receptor blockers (less than 24 hours before the sleep study).

Ages: 5 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children with and without sleep disorders, referred to Carmel Medical Center clinical sleep laboratory for an overnight sleep study
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2012-07; Primary Completion 2022-06 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Compare sleep data collected from the Watch-PAT device to PSG data | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Carmel Medical Center, Haifa, Israel